CLINICAL TRIAL: NCT06867068
Title: Comparison of Two Intravenous Drug Combinations for Ambulatory Oral & Maxillofacial Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2014-3556
Record Dates: First submitted 2025-03-05; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia; Tooth Extraction
Keywords: Ambulatory Oral Surgery; Maxillofacial Surgery; Intravenous; Ketamine; Propofol
MeSH Terms: interventions — Midazolam; Fentanyl; Ketamine; Propofol; Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: For purposes of safety the anesthesiologist was not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Group (Active Comparator): 1. Midazolam 0.05 mg/kg - rounded to closest ½ mg
  2. Fentanyl 50 micrograms (mcg) for patients less than or equal to 70kg and 75 mcg for those over 70 kg
  3. Ketamine 0.3 mg/kg - rounded to closest 5 mg (i.e., 70 kg patient - 3.5mg Midazolam, 50 mcg Fentanyl, 20 mg Ketamine)
  4. Additional intermittent dosage of Ketamine - 15 mg per surgeon's request
  All patients receive 40% nitrous oxide/oxygen, as per standard clinical care. All of the drugs are being used per label.
  Interventions: Drug: Midazolam Hydrochloride; Drug: Fentanyl; Drug: Ketamine; Drug: Nitrous oxide
- Propofol Group (Active Comparator): 1. Midazolam 0.05 mg/kg - rounded to closest ½ mg
  2. Fentanyl 50 mcg for patients less than or equal to 70 kg and 75 mcg for those over 70 kg
  3. Propofol 0.3 mg/kg - rounded to closest 5 mg (i.e., 70 kg patient - 3.5 mg Midazolam, 50 micrograms Fentanyl, 20 mg Propofol)
  4. Additional intermittent dosage of Propofol - 15 mg per surgeon's request
  All patients receive 40% nitrous oxide/oxygen, as per standard clinical care. All of the drugs are being used per label.
  Interventions: Drug: Midazolam Hydrochloride; Drug: Fentanyl; Drug: Propofol injection; Drug: Nitrous oxide

INTERVENTIONS:
Drug: Midazolam Hydrochloride — Short-acting sedative. Benzodiazepine. Gamma-aminobutyric acid (GABA) inhibitor
  Other Names: Versed
Drug: Fentanyl — Synthetic opioid drug used as an analgesic.
  Other Names: (N-phenyl-N-[1-(2-phenylethyl)-4piperidinyl]propanamide); Sublimaze, Actiq, Duragesic, Abstral, Subsys, and Ionsys
Drug: Ketamine — General Anesthetic. N-methyl-D-aspartate (NMDA) receptor agonist
  Other Names: Ketalar
  Arms: Ketamine Group
Drug: Propofol injection — General Anesthetic. GABA receptor modulator and calcium channel blocker
  Other Names: 2,6-diisopropylphenol; Diprivan
  Arms: Propofol Group
Drug: Nitrous oxide — Modulates a wide range of ligand-gated ion channels and inhibits NMDA receptor-mediated currents
  Other Names: Nitrous, laughing gas

SUMMARY:
The purpose of this pilot study was to compare two commonly employed intravenous drug combinations; I) nitrous oxide, midazolam, fentanyl, and ketamine and II) the same combination with substitution of propofol for ketamine, for use during wisdom teeth extraction. Measures of recovery, amnesia testing 20 minutes after induction and after completion of recovery tests, patient satisfaction, and surgeon satisfaction will be evaluated. The data from this pilot study will be used to obtain preliminary estimates of effect sizes and to select primary and secondary endpoints for the design of a larger scale and more definitive trial of the two anesthetic approaches.

DETAILED DESCRIPTION:
The widespread application of various ambulatory anesthetic techniques has paralleled the rapid rise of ambulatory surgery. It has been estimated that over half of all elective surgery is performed in an ambulatory setting. In addition, well over 3,000,000 intravenous sedations are administered in dental offices annually where local anesthesia is obtainable to control intraoperative pain. These intravenous sedation techniques have historically been an integral part of pain and anxiety control in the dental setting and have now gained widespread application in all of ambulatory surgery. A number of intravenous anesthetic techniques have been developed to achieve sedation levels ranging from conscious sedation where patients respond purposefully to verbal commands to deep sedation where patients cannot be easily aroused and protective reflexes may be altered. The goal of all of these techniques is to create a comfortable environment for the patient and a cooperative patient for the surgeon. Ideal technique should pose minimal physiologic challenge to the patient while providing amnesia for the procedure. Most of the intravenous sedation techniques in widespread use include a combination of drugs. These combinations function in an additive if not synergistic way. The pharmacological properties of their constituents achieve this ideal. The most frequently used drug when used alone and the most common to the various combinations is midazolam, a benzodiazepine. Midazolam has been shown to provide safe sedation with reliable anterograde amnesia. The duration of these effects is dose dependent. A short acting narcotic, usually fentanyl, is often times included to increase sedation levels and to add a modicum of analgesia. Other short acting agents can also be included to deepen the sedation level. These agents are usually added in incremental doses as the surgical setting requires. Both propofol and ketamine can induce general anesthesia but in significantly smaller doses provide additional sedation. These two agents come from different drug classes. Proponents of each cite advantages and disadvantages. Nitrous oxide is also commonly used in the dental setting.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) health class I or II
* Existing clinical population

Exclusion Criteria:

* Do not meet the Inclusion Criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | Postoperatively, approximately 1 hour on day of procedure
  Patient satisfaction was assessed using a patient evaluation survey administered following the procedure just prior to discharge. The survey consisted of 3 questions, 1 categorical and 2 ordinal. For purposes of this study, the 2 ordinal measures: "How do you feel now?" and "I would recommend this type of intravenous sedation to my family/friends" will be scored from 1-3 and 1-4, respectively for an overall possible scoring range of 2-7. Higher scores are associated with increased patient satisfaction. Satisfaction scores will be summarized by study arm.
Surgeon Satisfaction | Postoperatively, approximately 1 hour
  Surgeon satisfaction will be assessed by a surgeon's satisfaction survey administered following the procedure. The survey consisted of 3 questions which asked the surgeon to assess their level of satisfaction with the sedation regimen during local anesthesia, during the surgery, and overall satisfaction. Each of the three were rated as 1 ("Poor"), 2 ("Adequate"), or 3 ("Excellent") for an overall possible scoring range of 3-9. Higher scores are associated with increased surgeon satisfaction. Surgeon satisfaction scores will be summarized by study arm.
Recovery - Paper Test | Change from preoperatively to postoperatively, approximately 2-3 hours total on day of procedure
  Recovery will be assessed using a simple repeated measure paper and pencil test (PS Form 9a). This test presented participants with 25 rows of numbers. Each row consisted of a circled number at the beginning of the string of numbers. Patients were asked to cross out each number in a row that is like the circled number. The number of successfully completed rows were tabulated for each patient and change from baseline was summarized by study arm.
Recovery - One Leg Standing Test | Change from preoperatively to postoperatively, approximately 2-3 hours total on day of procedure
  Recovery will also be assessed by way of a 30 second one leg standing test administered prior to and following induction of anesthesia. The percentage of participants who are able to stand for at least 30 seconds will be summarized by study arm.
Amnesia - Visual Stimuli | Intraoperatively and postoperatively, up to 1-2 hours on day of procedure
  Amnesia will be evaluated by interrupting the procedure momentarily at specific intervals (approximately 20 minutes after induction and after completion of recovery test). Amnesia for visual stimuli will be assessed by having the patient verbally identify common objects (i.e., cup, pen, tape, and keys) presented during surgery. Patients will be asked to recall the items postoperatively. Recall of visual stimuli will be summarized by study arm using basic descriptive statistics.
Amnesia - Tactile Stimuli | Intraoperatively and postoperatively, up to 1-2 hours on day of procedure
  Amnesia will be evaluated by interrupting the procedure momentarily at specific intervals (approximately 20 minutes after induction and after completion of recovery test). Amnesia for tactile stimuli will be assessed by touching the patient with a pin on one of their four limbs and asking for recall. Recall of tactile stimuli will be summarized by study arm using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen S Gelfman, MD, DDS, Principal Investigator — New York City Health and Hospitals (NYCHHC)
Locations (1):
- NYCHHC - Jacobi Medical Center and North Central Bronx Hospital, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Association of Oral and Maxillofacial Surgeons Parameters of Care: Clinical Practice Guidelines. 2012.
- [Background] Braidy HF, Singh P, Ziccardi VB. Safety of deep sedation in an urban oral and maxillofacial surgery training program. J Oral Maxillofac Surg. 2011 Aug;69(8):2112-9. doi: 10.1016/j.joms.2011.04.017. PMID 21783001
- [Background] Craig DC, Wildsmith JA; Royal College of Anaesthetists; Royal College of Surgeons of England. Conscious sedation for dentistry: an update. Br Dent J. 2007 Dec 8;203(11):629-31. doi: 10.1038/bdj.2007.1105. PMID 18065980
- [Background] Goktay O, Satilmis T, Garip H, Gonul O, Goker K. A comparison of the effects of midazolam/fentanyl and midazolam/tramadol for conscious intravenous sedation during third molar extraction. J Oral Maxillofac Surg. 2011 Jun;69(6):1594-9. doi: 10.1016/j.joms.2010.09.005. Epub 2011 Feb 1. PMID 21277062
- [Background] Peskin RM. Contemporary intravenous anesthetic agents and delivery systems: propofol. Anesth Prog. 1992;39(4-5):178-84. No abstract available. PMID 1344020
- [Background] Sims PG, Kates CH, Moyer DJ, Rollert MK, Todd DW. Anesthesia in outpatient facilities. J Oral Maxillofac Surg. 2012 Nov;70(11 Suppl 3):e31-49. doi: 10.1016/j.joms.2012.07.030. No abstract available. PMID 23128005
- [Background] Ulmer BJ, Hansen JJ, Overley CA, Symms MR, Chadalawada V, Liangpunsakul S, Strahl E, Mendel AM, Rex DK. Propofol versus midazolam/fentanyl for outpatient colonoscopy: administration by nurses supervised by endoscopists. Clin Gastroenterol Hepatol. 2003 Nov;1(6):425-32. doi: 10.1016/s1542-3565(03)00226-x. PMID 15017641
- [Background] Personal Communication. Oral and Maxillofacial Surgery National Insurance Company. 2013.
- [Background] Blankstein KC. Low-dose intravenous ketamine: an effective adjunct to conventional deep conscious sedation. J Oral Maxillofac Surg. 2006 Apr;64(4):691-2. doi: 10.1016/j.joms.2005.11.038. No abstract available. PMID 16546650
- [Background] Casagrande AM. Propofol for office oral and maxillofacial anesthesia: the case against low-dose ketamine. J Oral Maxillofac Surg. 2006 Apr;64(4):693-5. doi: 10.1016/j.joms.2005.11.039. No abstract available. PMID 16546651
- [Background] Cillo JE Jr. Analysis of propofol and low-dose ketamine admixtures for adult outpatient dentoalveolar surgery: a prospective, randomized, positive-controlled clinical trial. J Oral Maxillofac Surg. 2012 Mar;70(3):537-46. doi: 10.1016/j.joms.2011.08.036. Epub 2011 Dec 16. PMID 22177821
- [Background] Driscoll EJ, Gelfman SS, Sweet JB, Butler DP, Wirdzck PR, Medlin T. Thrombophlebitis after intravenous use of anesthesia and sedation: its incidence and natural history. J Oral Surg. 1979 Nov;37(11):809-15. PMID 290773
- [Background] Haas DA, Harper DG. Ketamine: a review of its pharmacologic properties and use in ambulatory anesthesia. Anesth Prog. 1992;39(3):61-8. PMID 1308374
- [Background] Idvall J, Ahlgren I, Aronsen KR, Stenberg P. Ketamine infusions: pharmacokinetics and clinical effects. Br J Anaesth. 1979 Dec;51(12):1167-73. doi: 10.1093/bja/51.12.1167. PMID 526385
- [Background] Kramer KJ, Ganzberg S, Prior S, Rashid RG. Comparison of propofol-remifentanil versus propofol-ketamine deep sedation for third molar surgery. Anesth Prog. 2012 Fall;59(3):107-17. doi: 10.2344/12-00001.1. PMID 23050750
- [Background] Senel AC, Altintas NY, Senel FC, Pampu A, Tosun E, Ungor C, Dayisoylu EH, Tuzuner T. Evaluation of sedation in oral and maxillofacial surgery in ambulatory patients: failure and complications. Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 Nov;114(5):592-6. doi: 10.1016/j.oooo.2012.03.008. Epub 2012 Aug 15. PMID 22901639
- [Background] Gelfman SS, Gracely RH, Driscoll EJ, Wirdzek PR, Butler DP, Sweet JB. Comparison of recovery tests after intravenous sedation with diazepam-methohexital and diazepam-methohexital and fentanyl. J Oral Surg. 1979 Jun;37(6):391-7. PMID 286027
- [Background] Gelfman SS, Gracely RH, Driscoll EJ, Butler D, Sweet JB, Wirdzek PR. Recovery following intravenous sedation during dental surgery performed under local anesthesia. Anesth Analg. 1980 Oct;59(10):775-81. PMID 7191651
- [Background] Lepere AJ, Slack-Smith LM. Average recovery time from a standardized intravenous sedation protocol and standardized discharge criteria in the general dental practice setting. Anesth Prog. 2002 Summer;49(3):77-81. PMID 15384295
- [Background] Takarada T, Kawahara M, Irifune M, Endo C, Shimizu Y, Maeoka K, Tanaka C, Katayama S. Clinical recovery time from conscious sedation for dental outpatients. Anesth Prog. 2002 Winter;49(4):124-7. PMID 12779113
- [Background] Becker DE. Pharmacokinetic considerations for moderate and deep sedation. Anesth Prog. 2011 Fall;58(4):166-72; quiz 173. doi: 10.2344/0003-3006-58.4.166. PMID 22168806
- [Background] Gelfman SS, Gracely RH, Driscoll EJ, Wirdzek PR, Sweet JB, Butler DP. Conscious sedation with intravenous drugs: a study of amnesia. J Oral Surg. 1978 Mar;36(3):191-7. PMID 272450
- [Background] Miller RI, Bullard DE, Patrissi GA. Duration of amnesia associated with midazolam/fentanyl intravenous sedation. J Oral Maxillofac Surg. 1989 Feb;47(2):155-8. doi: 10.1016/s0278-2391(89)80108-9. PMID 2913250
- [Background] Bennett J, Peterson T, Burleson JA. Capnography and ventilatory assessment during ambulatory dentoalveolar surgery. J Oral Maxillofac Surg. 1997 Sep;55(9):921-5;discussion 925-6. doi: 10.1016/s0278-2391(97)90058-6. PMID 9294499
- [Background] Dionne RA, Driscoll EJ, Gelfman SS, Sweet JB, Butler DP, Wirdzek PR. Cardiovascular and respiratory response to intravenous diazepam, fentanyl, and methohexital in dental outpatients. J Oral Surg. 1981 May;39(5):343-9. PMID 6938649

DOCUMENTS (1):
  • Informed Consent Form (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT06867068/ICF_000.pdf